CLINICAL TRIAL: NCT05927311
Title: Prospective Study : Side Effects of Antibiotics in Bone and Joint Infections
Brief Title: Side Effects of Antibiotics in Bone and Joint Infections
Acronym: PROSEAB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR230121-PROSEAB
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Bone Infection; Joint Infection
Keywords: antibiotherapy; adverse events

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Treatment for bone and joint infection (BJI) is not standardized, which allows a wide range of antibiotic therapy to potentially be given, most often in high doses over long periods of time. Patients are regularly confronted with the adverse effects of these antibiotics, which can lead to loss of adherence and treatment failure. The frequency, severity and impact on quality of life of the adverse effects of long-term antibiotics will be studied in a cohort followed for one year.

DETAILED DESCRIPTION:
Treatment for bone and joint infection is not standardized, which allows a wide range of antibiotic therapy to potentially be given, most often in high doses over long periods of time. Patients are regularly confronted with the adverse effects of these antibiotics, which can lead to loss of adherence and treatment failure. Although patients with BJI receive regular follow-up, the impact of adverse events during treatments lasting more than a month is still poorly developed in the literature.

The frequency, severity and impact on quality of life of the adverse effects of long-term antibiotics will be studied in a cohort followed for one year.

The investigators believe that this study will improve the management of osteoarticular infections through a better understanding of the adverse effects associated with prolonged, high-dose antibiotic therapy, and encourage more multidisciplinary follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Microbiologically proven osteoarticular infection with or without material, requiring antibiotic therapy (single or multiple) of 6 weeks or more
* Oral antibiotic therapy (minimum 4 weeks)

Exclusion Criteria:

* Opposition to data processing
* Patient under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years of age with an osteoarticular infection requiring antibiotherapy of 6 weeks or more
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Adverse reactions | Day 15
  Changes in number, severity of clinical and biological adverse reactions to antibiotics reported by patients during follow-up of osteoarticular infections.
Adverse reactions | Day 45
  Changes in number, severity of clinical and biological adverse reactions to antibiotics reported by patients during follow-up of osteoarticular infections.
Adverse reactions | Day 90
  Changes in number, severity of clinical and biological adverse reactions to antibiotics reported by patients during follow-up of osteoarticular infections.

SECONDARY OUTCOMES:
Treatment failure | Day 15, day 45, day 90
  In the absence of the criterion of certainty, probable failure is defined by clinical (fever, pain, functional impotence, etc.), radiological (edging, signs of osteitis, etc.) and biological (increased CRP, hyperleukocytosis in the absence of any other cause) arguments.
compliance of treatment | Day 15, day 45, day 90
  Analysis of compliance and discontinuation of treatment, taking into account the adverse reaction profile.
Drug interactions | Day 15, day 45, day 90
  Analysis of drug interactions between antibiotic therapy for BJI and the patient's usual treatments at initiation and at each follow-up consultation.
EQ5D-5L | Day 365
  Quality of life will be assessed using the EuroQol 5 dimensions-5 levels (EQ-5D-5L) score questionnaire at the end of follow-up. Each one of the 5 scales goes from 1 to 5, 1 being the best possible outcome while 5 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Marion LACASSE, Principal Investigator — CHRU de Tours
Locations (1):
- University Hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided